CLINICAL TRIAL: NCT04539054
Title: Effects of a Multi-ingredient Pre-workout Supplement Versus Caffeine on Energy Expenditure and Feelings of Fatigue During Low-intensity Treadmill Exercise in College-aged Males.
Brief Title: Pre-workout Supplement Versus Caffeine on Energy Expenditure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Illinois University (Other)
Responsible Party: Principal Investigator, Clayton Camic, Associate Professor, Northern Illinois University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HS19-0163
Record Dates: First submitted 2020-08-26; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Healthy
Keywords: supplementation; ergogenic aid; metabolic rate; energy; substrate utilization

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-Workout Condition (Experimental): This condition consisted of the ingestion of one serving of the pre-workout supplement.
  Interventions: Dietary Supplement: ENGN Shred
- Caffeine Condition (Experimental): This condition consisted of the ingestion of 6 mg of caffeine per kg of body mass.
  Interventions: Dietary Supplement: Nutricost caffeine powder
- Placebo condition (Placebo Comparator): This condition consisted of the ingestion of a placebo.
  Interventions: Dietary Supplement: Crystal Light

INTERVENTIONS:
Dietary Supplement: ENGN Shred — ENGN Shred is a multi-ingredient pre-workout supplement.
  Arms: Pre-Workout Condition
Dietary Supplement: Nutricost caffeine powder — Caffeine powder.
  Arms: Caffeine Condition
Dietary Supplement: Crystal Light — Non-caloric Crystal Light matched for the pre-workout in terms of flavor and consistency.
  Arms: Placebo condition

SUMMARY:
The primary purpose of this study was to examine the acute effects of a multi-ingredient pre-workout supplement versus an ergogenic dose of caffeine (6 mg/kg) on energy expenditure during low-intensity exercise. The effects of these substances on substrate utilization, gas exchange, and psychological factors were also investigated. Twelve males (mean ± SD: age = 22.8 ± 2.4 years) completed three bouts of 60-min of treadmill exercise at 4.8-6.4 km/hr on separate days after consuming a pre-workout supplement, 6 mg/kg of caffeine, or placebo in a randomized fashion. The pre-workout and caffeine supplements resulted in significantly greater energy expenditure (p < 0.001, p = 0.006, respectively), VO2 (p < 0.001, p = 0.007, respectively), VCO2 (p = 0.006, p = 0.049, respectively), and VE (p < 0.001, p = 0.007, respectively), but not rates of fat or carbohydrate oxidation or respiratory exchange ratio compared to placebo (collapsed across condition). In addition, the pre-workout supplement increased feelings of alertness (p = 0.015) and focus (p = 0.005) 30-minutes post-ingestion and decreased feelings of fatigue (p = 0.014) during exercise compared to placebo (collapsed across condition). Thus, the pre-workout supplement increased energy expenditure and measures of gas exchange to the same extent as 6 mg/kg of caffeine with concomitant increased feelings of alertness and focus and decreased feelings of fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Male

Exclusion Criteria:

* history of medical or surgical events, including cardiovascular disease, metabolic, renal, hepatic, or musculoskeletal disorders;
* use of any medications
* use of nutritional supplements
* habitual use of caffeine (≥1 caffeinated beverage per day)
* participation in another clinical trial or investigation of another investigational product within 30 days prior to screening/enrollment.

Ages: 19 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Identify as male.
Enrollment: 12 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Energy expenditure | Measured continuously during 60 minutes of exercise for all three supplement conditions
  Measurement of caloric expenditure via gas exchange

SECONDARY OUTCOMES:
Oxygen consumption | Measured continuously during 60 minutes of exercise for all three supplement conditions
  Measurement of rate of oxygen consumption using a metabolic cart
Carbon dioxide production | Measured continuously during 60 minutes of exercise for all three supplement conditions
  Measurement of rate of carbon dioxide production using a metabolic cart
Minute ventilation | Measured continuously during 60 minutes of exercise for all three supplement conditions
  Measurement of ventilation rate using a metabolic cart
Feelings of fatigue | Baseline, 30-minutes post-ingestion of supplement, and at the 30-minute time point of exercise for all three supplement conditions
  Subjects were asked to rate their feelings of fatigue using a 5-point Likert scale
Feelings of energy | Baseline, 30-minutes post-ingestion of supplement, and at the 30-minute time point of exercise for all three supplement conditions
  Subjects were asked to rate their feelings of energy using a 5-point Likert scale
Feelings of focus | Baseline, 30-minutes post-ingestion of supplement, and at the 30-minute time point of exercise for all three supplement conditions
  Subjects were asked to rate their feelings of focus using a 5-point Likert scale
Feelings of alertness | Baseline, 30-minutes post-ingestion of supplement, and at the 30-minute time point of exercise for all three supplement conditions
  Subjects were asked to rate their feelings of focus using a 5-point Likert scale
Rate of fat oxidation | Measured continuously during 60 minutes of exercise for all three supplement conditions
  Fat oxidation was estimated thru measurements of gas exchange
Rate of carbohydrate oxidation | Measured continuously during 60 minutes of exercise for all three supplement conditions
  Carbohydrate oxidation was estimated thru measurements of gas exchange

CONTACTS AND LOCATIONS:
Overall Officials: Clayton L Camic, PhD, Principal Investigator — Northern Illinois University
Locations (1):
- Exercise Physiology Laboratory, DeKalb, Illinois, United States

IPD SHARING:
Plan to Share IPD: No